CLINICAL TRIAL: NCT04938934
Title: Factors That Determine the Responses to Meal Ingestion: Conditioning Effect of Previous Symptoms
Brief Title: Conditioning Effect of Previous Symptoms on the Responses to Meal Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR(AG)338/2016M
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-06

CONDITIONS: Healthy
Keywords: meal ingestion; postprandial responses; hedonic sensations; homeostatic sensations; Conditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aversive conditioning (Experimental)
  Interventions: Behavioral: Lipids infusion
- Sham conditioning (Sham Comparator)
  Interventions: Behavioral: Sham infusion

INTERVENTIONS:
Behavioral: Lipids infusion — Lipids infusion via intestinal tube
  Arms: Aversive conditioning
Behavioral: Sham infusion — Sham infusion via intestinal tube
  Arms: Sham conditioning

SUMMARY:
Meal ingestion induces sensations that are influenced by a series of conditioning factors.

Aim: to determine the conditioning effect of previous digestive symptoms to a standardized probe meal.

Controlled randomized parallel study in healthy subjects on the conditioning effect of previous digestive symptoms on the responses to a comfort meal. Digestive symptoms will be induced by lipid (or sham) infusion into the intestine. On three separate days, digestive sensations (satiety, abdominal bloating, digestive well-being, mood, discomfort) in response to a comfort meal will be measured before, during and after the intervention. Primary outcome: effect of conditioning on the sensation of digestive well-being measured by -5 to +5 scale after a comfort meal. Secondary aim: effect of conditioning on abdominal on homeostatic sensations (satiety, fullness, discomfort, nausea).

Participants (16 women, 8 in the intestinal infusion and 8 in the sham intervention) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the comfort meal will be administered 4 h after breakfast. Studies will be conducted in a quiet, isolated room. On each study day, participants will be intubated with a nasoduodenal feeding tube under fluoroscopic control for lipids or sham infusion. A comfort meal will be administered and perception of digestive sensations will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in digestive well-being in response to a comfort meal before and after conditioning. | 120 minutes
  Change in digestive well-being measured by a 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation) in response to a comfort meal before and after conditioning.

SECONDARY OUTCOMES:
Difference in fullness sensation in response to a comfort meal before and after conditioning | 120 minutes
  Change in fullness sensation by a 10 cm scale graded from 0 (not at all) to 10 (very much) in response to a comfort meal before and after conditioning.
Change in mood in response to a comfort meal before and after conditioning | 120 minutes
  Change in mood measured by a 10 cm scale graded from -5 (negative) to +5 (positive) in response to a comfort meal before and after conditioning.
Change in hunger/satiety in response to a comfort meal before and after conditioning | 120 minutes
  Change in mood measured by a 10 cm scale graded from -5 (extremely hungry) to +5 (completely satiate) in response to a comfort meal before and after conditioning
Change in discomfort in response to a comfort meal before and after conditioning | 120 minutes
  Change in the sensation of discomfort by a 10 cm scale graded from 0 (not at all) to 10 (very much) in response to a comfort meal before and after conditioning

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Livovsky DM, Pribic T, Azpiroz F. Food, Eating, and the Gastrointestinal Tract. Nutrients. 2020 Apr 2;12(4):986. doi: 10.3390/nu12040986. PMID 32252402
- [Background] Livovsky DM, Azpiroz F. Gastrointestinal Contributions to the Postprandial Experience. Nutrients. 2021 Mar 10;13(3):893. doi: 10.3390/nu13030893. PMID 33801924
- [Background] Livovsky DM, Barber C, Barba E, Accarino A, Azpiroz F. Abdominothoracic Postural Tone Influences the Sensations Induced by Meal Ingestion. Nutrients. 2021 Feb 18;13(2):658. doi: 10.3390/nu13020658. PMID 33670508
- [Derived] Nieto A, Livovsky DM, Azpiroz F. Conditioning by a Previous Experience Impairs the Rewarding Value of a Comfort Meal. Nutrients. 2023 May 9;15(10):2247. doi: 10.3390/nu15102247. PMID 37242129